CLINICAL TRIAL: NCT05518292
Title: Comparison of Analgesic Efficacy of Ultrasound Guided Rhomboid Intercostal Block Versus Serratus Anterior Plane Block for Mastectomy Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Nevert Adel, assist. prof. of anesthesia and pain management, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R.22.09.1830
Record Dates: First submitted 2022-08-13; First posted 2022-08-26 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rhomboid intercostal block (Active Comparator): Ultrasound guided RIB will apply with 10-12 MHz linear ultrasound transducer, in plane technique. Patients will placed in the sitting position. 22G spinal needle needle will be inserted to plane between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2 cm to 3 cm medially from the medial border of the scapula. 20 ml of bupivacaine 0.25% will inject into the fascial plane.
  Interventions: Other: rhomboid intercostal block
- serratus anterior plane block (Active Comparator): Patients will placed in the lateral position with the diseased side up. A 10-12 MHz linear ultrasound transducer is placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The fifth rib is identified in the mid-axillary line. The following muscles are identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). As an extra-reference point, the thoracodorsal artery is used to aid the identification of the plane superficial to the serratus muscle. The needle (22G spinal needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle. Under continuous ultrasound guidance, 20 ml of bupivacaine 0.25% will inject.
  Interventions: Other: serratus anterior plane block

INTERVENTIONS:
Other: rhomboid intercostal block — Ultrasound guided RIB will apply with 10-12 MHz linear ultrasound transducer, in plane technique. Patients will placed in the sitting position. 22G spinal needle needle will be inserted to plane between the rhomboid muscle and intercostal muscles over the T5-6 ribs 2 cm to 3 cm medially from the medial border of the scapula. 20 ml of bupivacaine 0.25% will inject into the fascial plane.
  Arms: rhomboid intercostal block
Other: serratus anterior plane block — Patients will placed in the lateral position with the diseased side up. A 10-12 MHz linear ultrasound transducer is placed over the mid-clavicular region of the thoracic cage in a sagittal plane. The fifth rib is identified in the mid-axillary line. The following muscles are identified easily overlying the fifth rib: the latissimus dorsi (superficial and posterior), teres major (superior) and serratus muscle (deep and inferior). As an extra-reference point, the thoracodorsal artery is used to aid the identification of the plane superficial to the serratus muscle. The needle (22G spinal needle) will be introduced in-plane with respect to the ultrasound probe targeting the plane superficial to the serratus muscle. Under continuous ultrasound guidance, 20 ml of bupivacaine 0.25% will inject.
  Arms: serratus anterior plane block

SUMMARY:
Breast surgeries are usually associated with sever postoperative pain ,good perioperative analgesic technique after breast surgery is always questionable .Thoracic epidural and paravertebral blocks became the gold standard techniques for pain relief ,however they may be associated with complications such as spinal cord injury, total spinal anesthesia ,inadvertent intravascular injection and pneumothorax . Recently , fascial plane blocks have been introduced as an alternative such as erector spinae plane block and serratus plane block Serratus plane block were introduced by Blanco et al where local anesthetic injected superficial to the muscle to provide nerve block of the lateral cutaneous branches of the intercostal nerves Rhomboid intercostal block is an interfascial plane block for chest wall analgesia, it was reported in 2016 as alternative to thoracic epidural and paravertebral blocks.

DETAILED DESCRIPTION:
This double blinded randomized(closed envelope technique) study will be conducted on eighty ASA I and II female patients aged between 20-60 years, undergoing modified radical mastectomy surgeries at Oncology Center Mansoura University (OCMU). The study will start at September 2022 and the recruitment will take approximately five months. The study duration can take about eight months. All patients undergoing general anesthesia. Informed consent will be taken after approval by the local ethics committee. The exclusion criteria included local skin infection , bleeding disorder ,coagulation abnormality ,spine or chest deformity , psychiatric disease, pregnancy and patients with allergy to any of the drug used .

Patients will be randomly assigned to either two groups according to the block used either rhomboid plane block in group R (n=30) received total volume of 20 ml of bupivacain 0.25% or serratus plane block group S (n=30) received total volume of 20 ml of bupivacaine 0.5% . The observer anesthetist and the surgeon were blinded to the solution. Operation will be performed by the same surgeon .Anesthetic management will be standardized and all patients will be premedicated with diazepam 5mg per orally at the morning of the surgery. Induction will be started with preoxygenation for 3 min, anesthesia will be induced with fentanyl (2ug/kg), 2 mg/kg propofol, muscle relaxation will be achieved by atracurium 0.05 mg kg and tracheal intubation will be achieved using suitable size of endotracheal tube . Anesthesia will be maintained with minimum alveolar concentration(MAC ) of isoflurane with air - oxygen and fentanyl 1µg/kg boluses and atracurium 0.2 mg/kg to maintain heart rate and pressure within 20% of their baseline values, the patients' lungs will be ventilated to maintain an ETCO2 of 30-35 mmHg. . Isoflurane will be discontinued at the start of skin closure, residual neuromuscular block will be antagonized with neostigmine 0.05 mg kg and atropine 0.025 mg kg and the trachea will be extubated. Heart rate ,end-tidal CO2, pulse oximetry and systolic blood pressure and diastolic blood pressure will be recorded before induction of anesthesia (baseline) and after induction of anesthesia then every 5min during surgery till end of surgery .

Post operative assessment:

In the PACU , patients were monitored for heart rate ,oxygen saturation ,systolic blood pressure and diastolic blood pressure for 1 hour postoperative by another anesthetist who was not aware of the study protocol . Patients were discharged to the surgical ward if they achieved score of 10 at modified Aldrete score .

Postoperative severity of pain which was assessed using VAS 1/2 hour after surgery, then at 1h, 2h, 4h, 6 h, 8h,12h and 24 h postoperatively . All patients were given IV ketorolac 30 mg/8 hour postoperatively and IV fentanyl 0.5µg/kg was available as rescue analgesia whenever VAS continued to be>40 mm after 30 min of ketorolac injection. Fentanyl injection could be repeated. The time for the first postoperative analgesic dose requirements and the total dose of 24hour postoperative fentanyl consumption were recorded . Postoperative nausea and vomiting (PONV) were assessed using a four-point numerical scale (0=no PONV, 1=mild nausea, 2=severe nausea or vomiting once, and 3=vomiting more than once), postoperative adverse effects and complications were recorded .

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II
* female patients
* aged between 20-60 years,
* undergoing modified radical mastectomy surgeries

Exclusion Criteria:

* local skin infection ,
* bleeding disorder ,
* coagulation abnormality ,
* spine or chest deformity ,
* psychiatric disease,
* pregnancy
* patients with allergy to any of the drug used

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
numerical analog score | half hour after finishing mastectomy
  0= no pain 10=sever pain
numerical analog score | 1 hour after finishing mastectomy
  0= no pain 10=sever pain
numerical analog score | 4 hour after finishing mastectomy
  0= no pain 10=sever pain
numerical analog score | 8 hour after finishing mastectomy
  0= no pain 10=sever pain
numerical analog score | 12 hour after finishing mastectomy
  0= no pain 10=sever pain
numerical analog score | 24 hour after finishing mastectomy
  0= no pain 10=sever pain

SECONDARY OUTCOMES:
required analgesia | half hour after mastectomy
  numerical analog score more than 4

CONTACTS AND LOCATIONS:
Locations (1):
- Yahya Wahba, Al Mansurah, Egypt